CLINICAL TRIAL: NCT03325257
Title: Two-years Follow-up of Melanoma Patients Treated by Nivolumab During the French ATU Program
Brief Title: Post-ATU Study of Nivolumab
Acronym: Post-ATU
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: RC17_0027
Record Dates: First submitted 2017-07-13; First posted 2017-10-30 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Melanoma
Keywords: Unresectable melanoma; metastatic melanoma; Immunotherapy; Nivolumab; Temporary Auhorization for Use (ATU)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Routine care — This study is an observational one - there is no change to the routine care. Patients received the Nivolumab independently of the study. Only data will be collected during this project.

SUMMARY:
Nivolumab obtained European Marketing authorization in June 2015. Before this date, a Temporary Authorization for Use (ATU) Program in France for nivolumab was set up between September 2014 and August 2015. This program enrolled approximately 600 melanoma patients (unresectable or metastatic).

It appears relevant to conduct a study on patients treated during the ATU to assess thoroughly patient characteristics, efficacy, safety, and patterns of use of nivolumab in real-life conditions.

DETAILED DESCRIPTION:
In order to reach goals of this study, collaboration had been established between BMS and the RIC-Mel network (network for Research and Clinical Investigational Research on Melanoma) (NCT03315468).

The RIC-Mel network has set up a national database in order to reference the active file of melanoma patients in France. The RIC-Mel database, supported by Nantes University Hospital, had been approved by French authorities (CCTIRS and CNIL). The RIC-Mel network is coordinated by Pr B. DRENO (Nantes University Hospital) and Pr C. LEBBE (Saint-Louis Hospital, AP-HP, Paris). Nowadays, 49 centres located all over the country are participating, with more than 19,000 melanoma patients included in the database. The RIC-Mel database is referred as one of the privileged access to any research program on melanoma by the Cancerology Group (GCC) of the French Society of Dermatology .

Based on this, BMS and the RIC-Mel network had established a partnership to set up a study in order to estimate the overall survival of melanoma patients treated by Nivolumab during the French ATU program.

Data are collected in the RIC-Mel database by participating centres. Information of centres, follow-up of activity, data reviewing and extractions are realized by the RIC-Mel network. Data analysis is performed by BMS following a developed statistical protocol.

Patients included in the study were patients with unresectable or advanced metastatic melanoma, which received at least one of Nivolumab, dispensed during the French ATU program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic melanoma cared in participating sites,
* Patients included in French nivolumab ATU program,
* Patients treated by at least one perfusion of nivolumab,
* Patients agreed to participate to the study.

Exclusion Criteria:

* Patients with unresectable or metastatic melanoma not included in French nivolumab ATU program,
* Patients having initiated Nivolumab after the 31th December 2015,
* Patients disagreed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival of patients included in the study thanks to subgroups of interest | 2 years
  Overall survival is defined as the time from index date (initiation of Nivolumab) until date of death due to any cause. Overall survival will be censored on the last date a subject was known to be alive. Estimates of survival rates will be realized for 1-year and 2-year survival. Median time will also be calculated.
  Subgroups of interest are described in the description of the first Secondary Outcome Measure.
  Safety Issue: No

SECONDARY OUTCOMES:
Distribution of melanoma patients included in the study in all subgroups of interest thanks to their clinical features at the time of treatment initiation | Day 1
  Subgroups of interest, based on information collected in medical records, were :
  * ECOG performance status (PF). ECOG PF is attempted to quantify cancer patients' general well-being and activities of daily life. The classifications were 0, 1 or ≥2.
  * LDH level. This level is considered as a prognostic factor: higher the LDH level, the worst the prognosis. The classifications were ≤Upper Limit of Normal (ULN), >ULN, >2 ULN or N/R (Unknown).
  * History of brain metastasis. These metastases are considered as one of the most difficult-to-treat complications of melanoma. The classifications were No or Yes.
  * Line of therapy. The classifications were 0, 1, 2 or >2.
  * BRAF status. BRAF is a proto-oncogene. Melanoma patients with BRAF mutation are eligible to targeted therapy.The classifications were Yes (mutated), No (wild-type) and Unknown (no research).
  * Number of metastatic sites. Safety Issue: No
Proportion of melanoma patients included in the study categorized by genders overall and by subgroups of interest | Day 1
  Distribution of females and males. This analyse will be performed for all the study population and by subgroups of interest (as defined in the primary Outcome Measure).Safety Issue: No
Distribution of age of melanoma patients included in the study overall and by subgroups of interest | Day 1
  Age of patients is the age at the start of Nivolumab treatment Safety Issue: No
Description of Nivolumab treatment of melanoma patients included in the study | 2 years
  Average and median of Nivolumab treatment duration and infusion number will be assessed. Median time to discontinuation, whatever the reason and median time to discontinuation of dose related to adverse events. Distribution of reasons for discontinuation.
  Safety Issue: No
Incidence of select grade 3, 4 and 5 adverse events (AE) in melanoma patients included in the study and related to Nivolumab treatment | 2 years
  An AE is defined as any undesirable experience or manifestation associated with the use of a medical product in a patient. AEs are categorized by grades, which refer to severity : Grade 3 - Severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated, disabling, limiting self-care activities of daily living, Grade 4 - Life-threatening consequences, urgent intervention indicated, Grade 5 - Death related to AE. Proportion of patients with at least one or more select AE, distribution, average and median time of AE occurrence, duration and evolution of AEs as well as description of action on Nivolumab treatment will also be assessed.
  Safety Issue: Yes
Progression-free survival of melanoma patients included in the study | 2 years
  Progression-free survival is defined as the time since Nivolumab initiation to either the first disease progression date or at last known tumour assessment date, or death due to any cause, whichever occurs first.
  Safety Issue: No
Objective response rate of melanoma patients included in the study | 2 years
  Objective response rate as the number of subjects with a best objective response of either a partial response of a complete response. Objective response rate is the proportion of patients with an objective response. Safety Issue: No

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte DRENO, PU-PH, Principal Investigator — Nantes University Hospital
Locations (17):
- France (17):
  - AP-HP Hôpital Ambroise Paré, Paris, Boulogne Billancourt
  - CHU de Grenoble, Grenoble, La Tronche
  - Chu Amiens, Amiens
  - Hopital St andré-CHU DE Bordeaux, Bordeaux
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu Dijon, Dijon
  - CH du Mans, Le Mans
  - Chru Lille, Lille
  - Centre Léon Bérard de Lyon, Lyon
  - Hospices Civils de Lyon: Lyon Sud, Lyon
  - Hôpitaux de Marseille, Marseille
  - CHU NICE, Nice
  - CH de PAU, Pau
  - CHU de Rouen, Rouen
  - Chu Toulouse, Toulouse
  - Ch Valence, Valence
  - Institut Gustave Roussy, Villejuif